CLINICAL TRIAL: NCT00718913
Title: A Phase II Trial of Postoperative Chemotherapy and Chemo-radiotherapy for Resected Adenocarcinoma of the Stomach and Gastro-esophageal Junction
Brief Title: Postoperative Chemotherapy and Chemo-radiotherapy for Resected Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.07
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer
Keywords: Adjuvant Gastric Cancer; Adjuvant chemotherapy; Adjuvant chemo-radiation; Capecitabine
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Cisplatin; Capecitabine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): TCX ->RT -> TCX
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Capecitabine; Radiation: Radiation

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be given at 60 mg/m2, as a 60-minute infusion every 3 weeks for 2 cycles before chemo-radiation. Four to five weeks after completion of chemo-radiation therapy, all patients will receive two more cycles of Docetaxel 60 mg/m2.
  Other Names: Taxotere
Drug: Cisplatin — Cisplatin will be given at 60 mg/m2, as 2-hour infusion every 3 weeks for 2 cycles before chemo-radiation. Four to five weeks after completion of chemo-radiation therapy, all patients will receive two more cycles of Cisplatin at 60 mg/m2.
  Other Names: CDDP
Drug: Capecitabine — Capecitabine will be given orally at 1800 mg/m2 days 1 through 14 divided in two daily doses before chemo-radiation. Four to five weeks after completion of chemo-radiation therapy, all patients will receive two more cycles of Capecitabine at 1800 mg/m2 days 1 through 14 (divided in two daily doses).
  Other Names: Xeloda
Radiation: Radiation — At the end of the second cycle of chemotherapy and one week of rest (day 27), a total of 45 Gy (1.8 Gy fx/d) of radiotherapy will be given.
  Other Names: RT
Drug: Capecitabine — Capecitabine will be administered orally during radiotherapy for radiosensitization(1650 mg/m2 per day divided in two daily doses, 5 days/week, on Monday through Friday).
  Other Names: Xeloda

SUMMARY:
This study will determine the feasibility of adjuvant chemotherapy and chemo-radiotherapy for patients with surgically resected adenocarcinoma of the stomach and gastro-esophageal junction.

DETAILED DESCRIPTION:
Patients with localized gastric cancer often relapse either locally or systemically. A strategy to reduce relapses at common sites would be beneficial. Our prior trial has proved the feasibility of administering FOLFIRI regimen as adjuvant chemotherapy combined with adjuvant chemoradiation in patients with excised with curative intend gastric cancer. It would be important to improve the treatment involving active regimen as adjuvant chemotherapy and optimizing chemoradiation by introducing capecitabine as a radiosensitizer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radically resected adenocarcinoma of the stomach and/or gastroesophageal junction with histologic proof of adenocarcinoma, pathologically staged T2-3, any N, M0
* No prior radiation therapy to the stomach or immunotherapy or chemotherapy for any reason
* Patients must have a life expectancy of at least 16 weeks and a performance status of < 2 ECOG scale
* Previous adjuvant chemotherapy with Irinotecan, Oxaliplatin and/or 5-FU based regimen. Patients who relapse within the first 6 months after the completion of adjuvant treatment are not eligible for the study.
* Patients must have adequate bone marrow function (defined as peripheral absolute granulocyte count of > 2.000/µL, and platelet count of > 100.000/µL), adequate liver function (bilirubin < 1,5 mg/dl), and adequate renal function (creatinine < 1,5 mg/dl
* Patients must be able to understand the nature of this study and give written informed consent

Exclusion Criteria:

* Patients with T1N0 carcinoma
* Positive cytology of pleural, or pericardial effusion or patients with any peritoneal disease diagnosed intra-operatively)
* Biopsy proof of lymph node metastases outside the study field such as supraclavicular, mediastinal, or para-aortic nodes
* Evidence of metastatic disease to distant organs
* Patients with cardiac disease graded as New York Heart Association Class III or IV, severe uncontrolled diabetes, hypertension, cerebron-vascular disease, or infection
* Patients with diabetic neuropathy
* Abnormalities of mental status such that either the patient cannot fully comprehend the therapeutic implications of the protocol or comply with the requirements
* Presence of concurrent or previous malignancies in the past 5 years (except for resected squamous or basal cell carcinoma of the skin)
* Pregnant women are excluded from study entry due to the teratogenic effects of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients completing protocol therapy (feasibility) | The feasibility will be defined as the proportion of patients who receive adjuvant chemotherapy and chemo-radiation over total registered

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment on each cycle
Toxicity profile | Toxicity assessment on each chemotherapy cycle
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Boukovinas, MD, Principal Investigator — "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology
Locations (8):
- Greece (8):
  - University Hospital of Crete Dept of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - General Hospital of Larissa Dept of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus